CLINICAL TRIAL: NCT05841407
Title: The Effect of Isotonic Beetroot Supplementation on High-intensity Time-trial Performance
Brief Title: Beetroot Supplementation and High Intensity Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Stephen Burns, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-2022-880
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Exercise Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both isotonic drinks (high nitrate or no nitrate) are deidentified and labelled (coded) by a third party not involved with the research. Randomisation is completed by a third party not involved in the testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High nitrate (Experimental): High nitrate isotonic drink
  Interventions: Dietary Supplement: High nitrate isotonic drink
- No nitrate (Active Comparator): No nitrate isotonic drink
  Interventions: Dietary Supplement: No nitrate isotonic drink

INTERVENTIONS:
Dietary Supplement: High nitrate isotonic drink — High nitrate (12.9 mmol) drink with carbohydrate and minerals
  Arms: High nitrate
Dietary Supplement: No nitrate isotonic drink — Carbohydrate and mineral isotonic drink
  Arms: No nitrate

SUMMARY:
Ingested beetroot contains inorganic nitrate which is later converted to nitric oxide (NO) in the bloodstream. NO is an important signaling molecule with several physiological functions in the body including acting as a vasodilator, expanding arteries and improving blood flow. Beetroot juice contain inorganic nitrate and consumption of beetroot has been shown to improve skeletal muscle contractility and metabolism enhancing high-intensity exercise performance. Isotonic sports drinks contain carbohydrates and sodium, which also improve exercise performance by providing exogenous glucose for energy to the working muscle and central nervous system and enabling faster absorption of fluid into the bloodstream. The ingestion of exogenous nitrate and isotonic-carbohydrate drink are recognized strategies for promoting exercise performance but whether they can be effectively combined has not been shown. This study will compare the salivary nitrite response, muscle oxygenation and time-trial performance after ingestion of two isotonic drinks with high in nitrate or with no nitrate.

DETAILED DESCRIPTION:
Ingested beetroot contains inorganic nitrate (NO3-) which is later converted to nitric oxide (NO) in the bloodstream. NO is an important signaling molecule with several physiological functions in the body including acting as a vasodilator, expanding arteries and improving blood flow. These functions mean that beetroot juice has become of strong interest in the field of exercise and is a recommended supplement for athletes to improve performance in recent consensus statements by the International Olympic Committee on dietary supplements. Importantly, the consumption of beetroot has been shown to improve skeletal muscle contractility and metabolism, hence, enhancing high-intensity exercise performance . Isotonic sports drinks contain carbohydrates and sodium, which also improve exercise performance by providing exogenous glucose for energy to the working muscle and central nervous system and enabling faster absorption of fluid into the bloodstream. The ingestion of exogenous nitrate and isotonic-carbohydrate drink are recognized strategies for promoting exercise performance but whether they can be effectively combined has not been shown. This study will compare the salivary nitrite response, muscle oxygenation and time-trial performance after ingestion of two drinks either high in nitrate or with no nitrate. Participants will ingest the two drinks in a randomised, crossover double-blind trial. One hour after drink ingestion they will undertake high intensity intermittent exercise for 30 minutes followed by a 10 km time trial on a cycle ergometer. Time trial will be compared between trials as the main outcome. It is hypothesised that the drink high in nitrate will lead to faster time trial completion.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 - 40 years
* Healthy and injury-free (e.g., no cardiovascular disease, diabetes mellitus, orthopaedic impairment that interferes with moderate-to-vigorous exercise)
* Blood pressure < 130/90 mmHg
* Physically active: Engaging in a minimum of 150 minutes of moderate-intensity exercise or 75 minutes of vigorous-intensity physical activity each week.
* Recreational cyclist (Minimum 1 hour cycling per week)
* Body mass index: 18.5-25 kg/m2
* Non-smoker
* Asian ethnicity by self identification

Exclusion Criteria:

* Any allergies to beetroot or isotonic drink.
* Asthma.
* Any report of personal health issues that may compromise the individual's ability to undertake exercise safely.
* Any recent Covid vaccination (within last 2 weeks).

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
10 km cycling time trial (endurance) performance | 1 hour after drink ingestion the time taken to complete 10 km on a stationary cycle ergometer will be assessed. Time to complete this is the primary outcome measure .
  Time trial

SECONDARY OUTCOMES:
Salivary nitrate | Four samples over 2 hours
  Salivary nitrate concentration determined from strips
Near infra-red spectroscopy (NIRS) | During cycling ~1 hour
  Tissue saturation index

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Burns, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Human Bioenergetics Laboratory, National Institute of Education, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All published data will be placed into the Data Repository of Nanyang Technological University National Institute of Education for public access upon publication.
Supporting Information: Analytic Code
Time Frame: Upon publication - permanent repository
Access Criteria: Public repository - exact web address available upon publication.
URL: http://researchdata.nie.edu.sg/